CLINICAL TRIAL: NCT01517347
Title: Low Dose of Interleukin-2 Following Allogeneic Unmanipulated Blood and Marrow Transplantation in Treating Patients With Standard Risk Hematologic Malignancy
Brief Title: Efficiency Study of Low Dose of IL-2 to Prevent Relapse in Standard Risk Leukemia After Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the conditional power was 0.083, the Data and Safety Monitoring Board recommended halting the study due to futility after the 1st interim analysis.
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, Chief of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUPH IRB [2012] (09）
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Leukemia
Keywords: IL2; relapse; GVHD; survival; allogeneic stem cell transplantation; MRD; CR
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin-2 (Experimental): Interleukin-2 post-transplantation to prevent relapse of standard risk leukemia
  Interventions: Drug: Interleukin-2
- controlled group (No Intervention): controlled standard risk leukemia received regular transplantation without IL-2 intervention

INTERVENTIONS:
Drug: Interleukin-2 — Patients receive low dose interleukin-2(Daily 1×106 IU per square meter of body-surface area) on days 60 after unmanipulated blood and marrow transplantation. Interleukin-2 treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: IL-2
  Arms: Interleukin-2

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is one of the best, and sometimes the only, option for the treatment of leukemia. However, relapse rate was still the key question to influence the overall survival after transplantation, even in standard risk leukemia.There were good evidences that natural killer cells and T regulatory cells, which were expanded and stimulated by the application of IL-2, could mediate protection against GvHD while maintaining graft anti-tumor activity as a positive side effect. Meanwhile, it was found in our previous pilot study that low-dose IL-2 subcutaneous administration from 100 days for a prolonged period could be a safe and effective strategy to prevent relapse in acute lymphoblastic malignancy patients with high risk of recurrence after unmanipulated allo-HSCT.

The study hypothesis:

Prevention of relapse using low dose IL-2 following hematopoietic stem cell transplantation in patients with standard risk acute leukemia can

* reduce relapse rate
* improve survival

DETAILED DESCRIPTION:
Standard risk patients over 15 years old(except Ph+ ALL, AML t(8;21) and T-ALL) undergone unmanipulated blood and marrow transplantation following day 60 post-transplantation were randomized into treated group (with low dose IL-2 treatment) or controlled group (without any intervention post-transplantation). The end points were safety and clinical and immunologic response.Following time is 24 months.

Primary Outcome Measures:

*To determine the feasibility and efficacy of administering an 6 course of subcutaneous IL-2 in this patient population. [ Time Frame: 2 years ]

Secondary Outcome Measures:

*To assess the immunologic impact of ultra-low dose subcutaneous IL-2 in patients after transplantation [ Time Frame: 2 years ] Estimated Enrollment:360 Study Start Date:Jan 2012 Estimated Study Completion Date:Jan 2016

Intervention Details Description:

*Drug: Interleukin-2 Dose will vary depending upon when participant enters the trial: Given as a daily injection under the skin for 8 weeks.

Detailed Description:

* Patients receive low dose interleukin-2(Daily 1×106 IU per square meter of body-surface area) on days 60 after unmanipulated blood and marrow transplantation. Interleukin-2 treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Participants will be seen periodically while they are receiving IL-2. Physical exams and blood tests will be performed weekly for the first two weeks and then every other week until the completion of 6 course therapy.

Eligibility Ages Eligible for Study:15 Years and older Genders Eligible for Study:Both Accepts Healthy Volunteers:No Criteria

Inclusion Criteria:

* Standard risk of Recipients of allogeneic stem cell transplantation with myeloablative conditioning regimens
* Standard risk of Recipients: CR1 or CR 2 of AML/ALL before transplantation
* Ph+ ALL，AML with t(8;21) and T-ALL were excepted
* Patients were at least 60 days post-transplantation
* Bone marrow monitoring was still Complete Remission (CR) and minor residual disease (MRD) was negative
* 15 years of age or older
* No serious infection

Exclusion Criteria:

* Exposure to any other clinical trials prior to enrollment
* Active malignant disease relapse
* Active, uncontrolled infection
* Inability to comply with IL-2 treatment regimen

ELIGIBILITY:
Inclusion Criteria:

* Standard risk of Recipients (CR1 or CR 2 of AML/ALL before transplantation except Ph+ ALL and T-ALL) of allogeneic stem cell transplantation with myeloablative conditioning regimens
* Standard risk of Recipients: CR1 or CR 2 of AML/ALL before transplantation
* Ph+ ALL, AML with t(8;21) and T-ALL were excepted
* Patients were at least 60 days post-transplantation
* Bone marrow monitoring was still Complete Remission (CR) and minor residual disease (MRD) was negative
* 15 years of age or older
* No serious infection

Exclusion Criteria:

* Exposure to any other clinical trials prior to enrollment
* Active malignant disease relapse
* Active, uncontrolled infection
* Inability to comply with IL-2 treatment regimen

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and efficiency of administering 6 courses of subcutaneous IL-2 in these patients population. | 2 years
  investigate the incidences of severe GVHD and pancytopenia after IL-2 application to evaluate the safety of this drug.
  observe the drug toxicity based on common toxicity criteria (CTC,version 3.0). compare the relapse rate and incidence of positive MRD between two groups to evaluate the efficiency of IL-2 application.

SECONDARY OUTCOMES:
To assess the immunologic impact of ultra-low dose subcutaneous IL-2 in patients after transplantation | 2 years
  examine the immune reconstitution of subgroups of T cells after IL-2 application and compare with that of controlled group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, MD, Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Xiaosu Zhao, Beijing, Beijing Municipality, China